CLINICAL TRIAL: NCT01211340
Title: The ACTIVE Intervention to Improve Hospice Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Debra Parker Oliver, Principle Investigator, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1160518
Record Dates: First submitted 2010-09-23; First posted 2010-09-29 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2017-04

CONDITIONS: Pain
Keywords: Hospice; Caregivers; Interdisciplinary Team; Pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Usual hospice care- there is no intervention in this arm
- ACTIVE (Experimental): Behavioral intervention using web conferencing
  Interventions: Behavioral: ACTIVE

INTERVENTIONS:
Behavioral: ACTIVE — Assessing Caregivers for Team Intervention via Video Encounters: this intervention uses video technology to bridge geographic distance to empower hospice caregivers to participate in plan of care meetings for their patient
  Arms: ACTIVE

SUMMARY:
The ACTIVE Intervention to Improve Hospice Caregiver Pain Management The major goal of this project is to implement and test this promising intervention in three hospice programs. The mixed methods evaluation of this randomized controlled trial (RCT) will provide evidence-based data for a tested intervention manual that hospice staff members can use to integrate the intervention into their practices.

DETAILED DESCRIPTION:
The ACTIVE Intervention to Improve Hospice Caregiver Pain Management The major goal of this project is to implement and test this promising intervention in three hospice programs. The mixed methods evaluation of this RCT will provide evidence-based data for a tested intervention manual that hospice staff members can use to integrate the intervention into their practices. We will rigorously test the effectiveness of the ACTIVE intervention. We will investigate whether the assessment of the informal caregivers perception of pain management will identify those who will benefit most and whether changes in the perceptions of informal caregivers will result in improvement of patient pain. We will explore barriers and challenges in the implementation of this into every day practice within hospice

ELIGIBILITY:
Inclusion Criteria: Informal Caregiver Inclusion Criteria

1. Informal caregiver of an enrolled hospice patient
2. Age 18 or over and legally able to provide informed consent
3. Involved in decisions related to pain medications
4. Access to at least one of the below:

   1. A standard land line telephone
   2. A high-speed Internet connection with operational computer
5. Without functional hearing loss or with a hearing aid that allows the participant to conduct phone or Internet conversations as assessed by the research staff (by questioning and observation

   -

   Exclusion Criteria:Informal caregivers of hospice patients with a life expectancy less than 14 days as assessed by the hospice nurse with the palliative performance scale (PPS) (99)

   -

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2010-09; Primary Completion 2014-04 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Parker Oliver, PhD, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - Hospice Compassus, Columbia, Missouri
  - Hands of Hope Hospice, Saint Joseph, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kruse RL, Parker Oliver D, Wittenberg-Lyles E, Demiris G. Conducting the ACTIVE randomized trial in hospice care: keys to success. Clin Trials. 2013 Feb;10(1):160-9. doi: 10.1177/1740774512461858. Epub 2012 Oct 25. PMID 23104974
- [Result] Parker Oliver D, Demiris G, Washington K, Kruse RL, Petroski G. Hospice Family Caregiver Involvement in Care Plan Meetings: A Mixed-Methods Randomized Controlled Trial. Am J Hosp Palliat Care. 2017 Nov;34(9):849-859. doi: 10.1177/1049909116661816. Epub 2016 Jul 27. PMID 27465403
- [Derived] Washington KT, Demiris G, Pike KC, Kruse RL, Oliver DP. Anxiety among informal hospice caregivers: an exploratory study. Palliat Support Care. 2015 Jun;13(3):567-73. doi: 10.1017/S1478951513001193. Epub 2014 Feb 13. PMID 24524662
- [Derived] Parker Oliver D, Albright DL, Washington K, Wittenberg-Lyles E, Gage A, Mooney M, Demiris G. Hospice caregiver depression: the evidence surrounding the greatest pain of all. J Soc Work End Life Palliat Care. 2013;9(4):256-71. doi: 10.1080/15524256.2013.846891. PMID 24295096
- [Derived] Albright DL, Kruse RL, Oliver DP, Washington K, Cagle J, Demiris G. Testing the factorial validity of scores from the caregiver pain medicine questionnaire. J Pain Symptom Manage. 2014 Jul;48(1):99-109. doi: 10.1016/j.jpainsymman.2013.08.014. Epub 2013 Nov 15. PMID 24246789
- [Derived] Wittenberg-Lyles E, Goldsmith J, Oliver DP, Demiris G, Kruse RL, Van Stee S. Using medical words with family caregivers. J Palliat Med. 2013 Sep;16(9):1135-9. doi: 10.1089/jpm.2013.0041. Epub 2013 Aug 12. PMID 23937064
- [Derived] Demiris G, Parker Oliver D, Capurro D, Wittenberg-Lyles E. Implementation science: implications for intervention research in hospice and palliative care. Gerontologist. 2014 Apr;54(2):163-71. doi: 10.1093/geront/gnt022. Epub 2013 Apr 4. PMID 23558847
- [Derived] Wittenberg-Lyles E, Goldsmith J, Oliver DP, Demiris G, Kruse RL, Van Stee S. Exploring oral literacy in communication with hospice caregivers. J Pain Symptom Manage. 2013 Nov;46(5):731-6. doi: 10.1016/j.jpainsymman.2012.11.006. Epub 2013 Mar 21. PMID 23522518
- [Derived] Baldwin PK, Wittenberg-Lyles E, Kruse RL, Demiris G, Parker Oliver D. Pain management and the African American hospice caregiver: a case report. Am J Hosp Palliat Care. 2013 Dec;30(8):795-8. doi: 10.1177/1049909112469274. Epub 2012 Dec 10. No abstract available. PMID 23233538
- [Derived] Washington KT, Wittenberg-Lyles E, Parker Oliver D, Demiris G, Shaunfield S, Crumb E. Application of the VALUE communication principles in ACTIVE hospice team meetings. J Palliat Med. 2013 Jan;16(1):60-6. doi: 10.1089/jpm.2012.0229. Epub 2012 Oct 4. PMID 23036014

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: This arm serves as the control, individuals will not receive the intervention but will receive all measures
- Intervention Arm: These caregivers will receive usual care plus the technology which allows them to participate in their plan of care meeting
  ACTIVE: Assessing Caregivers for Team Intervention via Video Encounters: this intervention uses video technology to bridge geographic distance to empower hospice caregivers to participate in plan of care meetings for their patient
Period: Overall Study
Arm/Group | Usual Care | Intervention Arm
Started | 223 | 223
Completed | 223 | 223
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention Arm | Total
Number analyzed (Participants) | 223 | 223 | 446
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (13.3) | 60.1 (12.5) | 59.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 168 | 350
  Male | 41 | 55 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 221 | 220 | 441
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 7 | 9
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 10 | 23
  White | 205 | 204 | 409
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 223 | 223 | 446

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Perceptions of Pain Medicine Questionaire
Description: This 16 question instrument measures the perceptions hospice caregivers have toward the administration of pain medications. Scores on items vary from 1-5 with the lower scores indicating more problematic perceptions of pain management. A Total score is computed between 16-80 Only the last available measure will be used to reflect the measure closest to time of death.
Time Frame: Every 14 days until the death of the patient for an average of 45 days-Only measure used in analysis is the last completed measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention Arm
Number analyzed (Participants) | 223 | 223
units on a scale
  Baseline | 49.6 (7.3) | 49 (7.43)
  Last Measure | 50.3 (7.12) | 50.5 (7.33)
Statistical Analysis 1: Comparison: Usual Care vs Intervention Arm; The first analysis examined change from baseline to last available measure prior to death or the end of the study. The pre/post change was calculated for each participant and the Wilcoxon rank sum test was used to compare usual care and intervention groups with respect to changes. All randomized caregivers with at least 1 post baseline measure were included in the analysis; Test type: Superiority or Other; p = .18, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Usual Care vs Intervention Arm; The secondary analysis used a linear mixed model to test for groups differences over time. To account for repeated- measures nature of the data and the varying duration of participation, both participant specific intercept and slopes were treated as random effects. To minimize the leverage of relatively small number of participants with extremely long follow-up times we limited the number of days followed to 122, which was the 75th percentile of the days in the combined study; Test type: Superiority or Other; p = .18, Regression, Linear; No significant difference found between groups
Statistical Analysis 3: Comparison: Usual Care vs Intervention Arm; To test the effects of the dose of meetings on association with overall Caregiver Perceptions of Pain Medicine Questionaire (CPMQ) change we used Spearman rank correlation coefficient; Test type: Superiority or Other; p = .18, Spearmans rank; No differences found

2. Secondary Outcome: Caregiver Quality of Life-Revised Subscale Emotional
Description: This is one domain of a four domain instrument. It involves one question with a range of 0-10.Only the last available measure will be used to reflect the measure closest to time of death.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention Arm
Number analyzed (Participants) | 223 | 223
units on a scale
  Baseline | 7.06 (2.26) | 7.61 (1.93)
  Last Measure | 6.95 (2.08) | 7.19 (2.03)
Statistical Analysis 1: Comparison: Usual Care vs Intervention Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .15, Wilcxon Rank Sum Test
Statistical Analysis 2: Comparison: Usual Care vs Intervention Arm; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = .15, Regression, Linear

3. Secondary Outcome: Anxiety
Description: This measure determines the level of anxiety experienced by a hospice caregiver. Total scores range from 0-21 with higher scores representing more anxiety. Only the last available measure will be used to reflect the measure closest to time of death.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention Arm
Number analyzed (Participants) | 223 | 223
units on a scale
  Baseline | 6.65 (5.33) | 5.86 (5.16)
  Last Measure | 6.37 (5.81) | 5.86 (5.16)
Statistical Analysis 1: Comparison: Usual Care vs Intervention Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .89, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Usual Care vs Intervention Arm; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = .89, Regression, Linear

ADVERSE EVENTS:
Arm/Group | Usual Care | Intervention Arm
Serious Adverse Events (participants affected / at risk) | 0/223 | 0/223
Other Adverse Events (participants affected / at risk) | 0/223 | 0/223

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No